CLINICAL TRIAL: NCT00601731
Title: A Phase 2, Open-label, Controlled, Multi-center Study to Evaluate Meningococcal ACWY Antibody Response in Children Aged 40 and 60 Months Who Have Previously Received Novartis MenACWY Conjugate Vaccine as Infants
Brief Title: Evaluation of Meningococcal ACWY Immune Response in Children Aged 40 and 60 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P5E1; 2007-004978-16
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Meningococcal Disease
Keywords: Prevention of Meningococcal disease
MeSH Terms: conditions — Meningococcal Infections | interventions — Hematologic Tests

ARMS (2):
- Adjuvanted MenACWY vaccine group (Experimental): Blood test
  Interventions: Biological: MenACWY-CRM197
- Non-adjuvanted MenACWY vaccine group (Active Comparator): Blood test
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: MenACWY-CRM197 — Blood test, 40-months and 60-months children
  Arms: Adjuvanted MenACWY vaccine group
Biological: Blood test — Blood test, 40-months and 60-months children
  Arms: Non-adjuvanted MenACWY vaccine group

SUMMARY:
The purpose of this study is to evaluate how well the immuno response against meningococcal serogroups A, C, W and Y lasts in children who were vaccinated with MenACWY as infants.

ELIGIBILITY:
Inclusion Criteria:

* Follow-on, healthy 40, 60 months old participants who have completed the V59P5 study and are in good health
* Control subjects: healthy 60 months old who had received a complete MenC immunization course

Exclusion Criteria:

* Subjects with any serious, acute or chronic progressive disease

Ages: 40 Months to 63 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 382 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- Canada (2):
  - Clinical Trials Research Center, Halifax
  - Vaccine Evaluation Center, Vancouver
- Oxford Vaccine Group, Oxford, United Kingdom

REFERENCES:
- [Derived] Khatami A, Snape MD, Davis E, Layton H, John T, Yu LM, Dull PM, Gill CJ, Odrjlin T, Dobson S, Halperin SA, Langley JM, McNeil SA, Pollard AJ. Persistence of the immune response at 5 years of age following infant immunisation with investigational quadrivalent MenACWY conjugate vaccine formulations. Vaccine. 2012 Apr 16;30(18):2831-8. doi: 10.1016/j.vaccine.2012.02.046. Epub 2012 Mar 3. PMID 22394992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 3 sites (1 site in the UK and 2 sites in Canada).
Groups:
- UK Site: UK vaccine group that received primary vaccine schedule of MenACWY (adjuvanted and unadjuvanted) vaccine at 2, 3 and 4 months with booster at 12 months of age, enrolled at either 40 or 60 months of age into the current study as follow-on participants.
- UK Control: Newly enrolled age-matched subjects that received a complete vaccination course of routine monovalent MenC conjugate vaccine at 2, 3 and 4 months of age without any booster vaccination.
- Canada Sites: Canadian vaccine group that received primary vaccination with MenACWY (adjuvanted and unadjuvanted) vaccine at 2,4 months of age with 12 month booster or at 2, 4, 6 months with or without a booster vaccination.
- Canada Control: Newly enrolled age-matched subjects that received the complete vaccination course of routine monovalent MenC conjugate vaccine at 2 and 12 months or only at 12 months of age.
Period: Overall Study
Arm/Group | UK Site | UK Control | Canada Sites | Canada Control
Started | 143 | 43 | 166 | 30
Completed | 120 | 43 | 151 | 29
Not Completed | 23 | 0 | 15 | 1

BASELINE CHARACTERISTICS:
Groups:
- UK2,3,4,12+: UK vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 2, 3, and 4 months of age followed by a booster dose of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 12 months of age.
- UK2,4,12+: UK vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 2 and 4 months of age followed by a booster dose of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 12 months of age.
- UK2,4C/12+: UK vaccine group receiving primary vaccine of monovalent MenC-CRM197 conjugate vaccine (Menjugate) at 2 and 4 months of age followed by a booster dose of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 12 months of age.
- UK2,4,12-: UK vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine without adjuvant at 2 and 4 months of age followed by a booster dose of quadrivalent MenACWY-CRM197 conjugate vaccine without adjuvant at 12 months of age.
- Ca2,4,6+: Canadian vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 2, 4 and 6 months of age without any booster vaccination.
- Ca2,4,6+/12PS: Canadian vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 2, 4 and 6 months of age followed by a reduced booster vaccination of quadrivalent MenACWY polysaccharide vaccine (Menomune [1/5 dose]) at 12 months of age
- Ca2,4,12+: Canadian vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 2 and 4 months of age followed by a booster dose of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 12 months of age.
- Ca2,4+/12PS: Canadian vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine with adjuvant at 2 and 4 months of age followed by a reduced booster vaccination of quadrivalent MenACWY polysaccharide vaccine (Menomune [1/5 dose]) at 12 months of age.
- Ca2,4,12-: Canadian vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine without adjuvant at 2 and 4 months of age followed by a booster vaccination of the quadrivalent MenACWY-CRM197 conjugate vaccine without adjuvant at 12 months of age.
- Ca2,4-/12PS: Canadian vaccine group receiving primary vaccine of quadrivalent MenACWY-CRM197 conjugate vaccine without adjuvant at 2 and 4 months of age followed by a reduced booster vaccination of the quadrivalent MenACWY polysaccharide vaccine (Menomune [1/5 dose]) at 12 months of age.
- Ca Control: Newly enrolled age-matched subjects that received a complete vaccination course of routine monovalent MenC conjugate vaccine at 2 and 12 months or only at 12 months of age.
- Total: Total of all reporting groups
Arm/Group | UK2,3,4,12+ | UK2,4,12+ | UK2,4C/12+ | UK2,4,12- | UK Control | Ca2,4,6+ | Ca2,4,6+/12PS | Ca2,4,12+ | Ca2,4+/12PS | Ca2,4,12- | Ca2,4-/12PS | Ca Control | Total
Number analyzed (Participants) | 40 | 44 | 22 | 37 | 43 | 31 | 26 | 27 | 28 | 27 | 27 | 30 | 382
Age, Customized [Mean (Standard Deviation); unit: months]
  40 months (N=36,37,19,34,0,28,23,27,28,25,26,0) | 42.4 (0.7) | 42.6 (0.6) | 42.6 (0.5) | 40.6 (0.8) | NA (NA) — Zero participants were in this subgroup. | 42 (1) | 41.8 (1.2) | 42 (0.9) | 41.6 (1) | 40.7 (1) | 41.0 (1.1) | NA (NA) — Zero participants were in this subgroup. | 34.78 (0.31)
  60 months (N=4,7,3,3,43,3,3,0,0,2,1,30) | 61.3 (1.0) | 61.3 (0.5) | 61.0 (1.0) | 61.7 (0.6) | 61.9 (0.3) | 60.3 (0.6) | 61.3 (0.6) | NA (NA) — Zero participants in this subgroup. | NA (NA) — Zero participants in this subgroup. | 60.5 (0.7) | 60.0 (0.0) | 60.6 (0.6) | 60.88 (0.16)
Sex/Gender, Customized [Number; unit: Number of subjects]
  Female 40 months | 14 | 19 | 14 | 19 | NA — Zero participants were in this subgroup. | 19 | 9 | 15 | 10 | 12 | 14 | NA — Zero participants were in this subgroup. | 145
  Male 40 months | 22 | 18 | 5 | 15 | NA — Zero participants were in this subgroup. | 9 | 14 | 12 | 18 | 13 | 12 | NA — Zero participants were in this subgroup. | 138
  Female 60 months | 1 | 4 | 1 | 2 | 20 | 2 | 3 | NA — Zero participants in this subgroup. | NA — Zero participants in this subgroup. | 1 | 0 | 15 | 49
  Male 60 months | 3 | 3 | 2 | 1 | 23 | 1 | 0 | NA — Zero participants in this subgroup. | NA — Zero participants in this subgroup. | 1 | 1 | 15 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With hSBA ≥1:8
Description: Percentages of subjects with human Serum Bactericidal Assay (hSBA) ≥1:8 as measured by serum bactericidal activity at 40 months and 60 months of age and associated 95% Clopper-Pearson CIs were computed for each of the serogroups within each of the vaccinated groups and in age-matched control subjects.
Time Frame: At 40 and 60 months of age
Population: Immunogenicity was evaluated in the Modified Intent To Treat (MITT) population that included subjects who provided at least one evaluable blood sample. Thus, the difference in the number of subjects entered here versus the number of subjects in the participant flow and baseline characteristics (i.e., enrolled subjects) module.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | UK2,3,4,12+ | UK2,4,12+ | UK2,4C/12+ | UK2,4,12- | UK Control | Ca2,4,6+ | Ca2,4,6+/12PS | Ca2,4,12+ | Ca2,4+/12PS | Ca2,4,12- | Ca2,4-/12PS | Ca Control
Number analyzed (Participants) | 33 | 37 | 18 | 34 | 42 | 28 | 25 | 27 | 28 | 25 | 24 | 30
Percentages of subjects
  MenA 40mths N=33,37,17,34,0,28,23,27,28,25,24,0 | 27 [13 to 46] | 8 [2 to 22] | 29 [10 to 56] | 3 [0.074 to 15] | NA [NA to NA] — zero participants analyzed | 0 [0 to 12] | 4 [0 to 22] | 7 [1 to 24] | 0 [0 to 12] | 8 [1 to 26] | 0 [0 to 14] | NA [NA to NA] — zero participants analyzed
  MenA 60mths N=33,35,18,31,42,27,25,23,25,23,24,30 | 9 [2 to 24] | 11 [3 to 27] | 11 [1 to 35] | 3 [0.082 to 17] | 0 [0 to 8] | 0 [0 to 13] | 0 [0 to 14] | 4 [0 to 22] | 4 [0 to 20] | 4 [0 to 22] | 0 [0 to 14] | 3 [0.084 to 17]
  MenC 40mths N=32,36,17,33,0,20,22,26,26,24,24,0 | 41 [24 to 59] | 47 [30 to 65] | 71 [44 to 90] | 33 [18 to 52] | NA [NA to NA] — zero participants analyzed | 20 [6 to 44] | 14 [3 to 35] | 31 [14 to 52] | 35 [17 to 56] | 38 [19 to 59] | 46 [26 to 67] | NA [NA to NA] — zero participants analyzed
  MenC 60mths N=32,34,17,31,42,21,24,22,21,22,24,30 | 34 [19 to 53] | 32 [17 to 51] | 59 [33 to 82] | 45 [27 to 64] | 29 [16 to 45] | 14 [3 to 36] | 13 [3 to 32] | 14 [3 to 35] | 24 [8 to 47] | 27 [11 to 50] | 46 [26 to 67] | 53 [34 to 72]
  MenW 40mths N=33,36,17,34,0,28,23,27,28,25,24,0 | 73 [54 to 87] | 69 [52 to 84] | 71 [44 to 90] | 74 [56 to 87] | NA [NA to NA] — zero participants analyzed | 29 [13 to 49] | 48 [27 to 69] | 59 [39 to 78] | 43 [24 to 63] | 72 [51 to 88] | 58 [37 to 78] | NA [NA to NA] — zero participants analyzed
  MenW 60mths N=32,34,18,31,42,26,25,23,24,21,24,29 | 69 [50 to 84] | 85 [69 to 95] | 78 [52 to 94] | 84 [66 to 95] | 36 [22 to 52] | 31 [14 to 52] | 44 [24 to 65] | 57 [34 to 77] | 42 [22 to 63] | 81 [58 to 95] | 67 [45 to 84] | 34 [18 to 54]
  MenY 40mths N=33,36,17,34,0,28,23,27,28,25,24,0 | 76 [58 to 89] | 61 [43 to 77] | 76 [50 to 93] | 53 [35 to 70] | NA [NA to NA] — zero participants analyzed | 32 [16 to 52] | 26 [10 to 48] | 44 [25 to 65] | 21 [8 to 41] | 64 [43 to 82] | 63 [41 to 81] | NA [NA to NA] — zero participants analyzed
  MenY 60mths N=33,34,17,31,42,27,25,23,23,21,23,30 | 61 [42 to 77] | 71 [53 to 85] | 71 [44 to 90] | 42 [25 to 61] | 29 [16 to 45] | 30 [14 to 50] | 24 [9 to 45] | 43 [23 to 66] | 22 [7 to 44] | 57 [34 to 78] | 57 [34 to 77] | 10 [2 to 27]

2. Secondary Outcome: Percentage of Subjects With hSBA ≥1:4
Description: Percentages of subjects with hSBA ≥1:4 as measured by serum bactericidal activity at 40 months and 60 months of age and associated 95% Clopper-Pearson CIs were computed for each of the serogroups within each of the vaccinated groups and in age-matched control subjects.
Time Frame: At 40 and 60 months of age
Population: The analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | UK2,3,4,12+ | UK2,4,12+ | UK2,4C/12+ | UK2,4,12- | UK Control | Ca2,4,6+ | Ca2,4,6+/12PS | Ca2,4,12+ | Ca2,4+/12PS | Ca2,4,12- | Ca2,4-/12PS | Ca Control
Number analyzed (Participants) | 33 | 37 | 18 | 34 | 42 | 28 | 25 | 27 | 28 | 25 | 24 | 30
Percentages of subjects
  MenA 40mths N=33,37,17,34,0,28,23,27,28,25,24,0 | 30 [16 to 49] | 8 [2 to 22] | 29 [10 to 56] | 3 [0.074 to 15] | NA [NA to NA] — Zero participants analyzed | 0 [0 to 12] | 4 [0 to 22] | 11 [2 to 29] | 7 [1 to 24] | 8 [1 to 26] | 0 [0 to 14] | NA [NA to NA] — Zero participants analyzed
  MenA 60mths N=33,35,18,31,42,27,25,23,25,23,24,30 | 15 [5 to 32] | 11 [3 to 27] | 22 [6 to 48] | 3 [0.082 to 17] | 0 [0 to 8] | 4 [0.094 to 19] | 0 [0 to 14] | 9 [1 to 28] | 4 [0 to 20] | 9 [1 to 28] | 0 [0 to 14] | 7 [1 to 22]
  MenC 40mths N=32,36,17,33,0,20,22,26,26,24,24,0 | 47 [29 to 65] | 53 [35 to 70] | 71 [44 to 90] | 42 [25 to 61] | NA [NA to NA] — Zero participants analyzed | 20 [6 to 44] | 14 [3 to 35] | 38 [20 to 59] | 54 [33 to 73] | 54 [33 to 74] | 54 [33 to 74] | NA [NA to NA] — Zero participants analyzed
  MenC 60mths N=32,34,17,31,42,21,24,22,21,22,24,30 | 50 [32 to 68] | 44 [27 to 62] | 71 [44 to 90] | 52 [33 to 70] | 40 [26 to 57] | 24 [8 to 47] | 29 [13 to 51] | 32 [14 to 55] | 48 [26 to 70] | 59 [36 to 79] | 58 [37 to 78] | 67 [47 to 83]
  MenW 40mths N=33,36,17,34,0,28,23,27,28,25,24,0 | 73 [54 to 87] | 69 [52 to 84] | 71 [44 to 90] | 85 [69 to 95] | NA [NA to NA] — Zero participants analyzed | 29 [13 to 49] | 52 [31 to 73] | 63 [42 to 81] | 54 [34 to 72] | 72 [51 to 88] | 71 [49 to 87] | NA [NA to NA] — Zero participants analyzed
  MenW 60mths N=32,34,18,31,42,26,25,23,24,21,24,29 | 69 [50 to 84] | 85 [69 to 95] | 83 [59 to 96] | 84 [66 to 95] | 39 [22 to 52] | 31 [14 to 52] | 52 [31 to 72] | 61 [39 to 80] | 50 [29 to 71] | 81 [58 to 95] | 67 [45 to 84] | 34 [18 to 54]
  MenY 40mths N=33,36,17,34,0,28,23,27,28,25,24,0 | 76 [58 to 89] | 78 [61 to 90] | 88 [64 to 99] | 71 [53 to 85] | NA [NA to NA] — Zero participants analyzed | 50 [31 to 69] | 35 [16 to 57] | 59 [39 to 78] | 43 [24 to 63] | 68 [46 to 85] | 63 [41 to 81] | NA [NA to NA] — Zero participants analyzed
  MenY 60mths N=33,34,17,31,42,27,25,23,23,21,23,30 | 73 [54 to 87] | 79 [62 to 91] | 76 [50 to 93] | 55 [36 to 73] | 33 [20 to 50] | 48 [29 to 68] | 40 [21 to 61] | 57 [34 to 77] | 35 [16 to 57] | 62 [38 to 82] | 61 [39 to 80] | 13 [4 to 31]

3. Secondary Outcome: GMTs in Subjects Within Each Site and in Age-Matched Control Subjects
Description: The Geometric Mean Titers (GMTs) as measured by serum bactericidal activity at 40 months and 60 months of age and 95% CIs were calculated for each vaccine group and for each serogroup by exponentiating (base 10) the least square means of the logarithmically transformed (base 10) titers and their 95% CIs obtained from a two-way Analysis of Variance (ANOVA) with factors for vaccine group and center.
Time Frame: At 40 and 60 months of age
Population: The analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | UK2,3,4,12+ | UK2,4,12+ | UK2,4C/12+ | UK2,4,12- | UK Control | Ca2,4,6+ | Ca2,4,6+/12PS | Ca2,4,12+ | Ca2,4+/12PS | Ca2,4,12- | Ca2,4-/12PS | Ca Control
Number analyzed (Participants) | 33 | 37 | 18 | 34 | 42 | 28 | 25 | 27 | 28 | 25 | 24 | 30
Titers
  MenA 40mths N=33,37,17,34,0,28,23,27,28,25,24,0 | 3.75 [2.76 to 5.11] | 2.58 [1.93 to 3.45] | 4.33 [2.82 to 6.66] | 2.08 [1.54 to 2.82] | NA [NA to NA] — Zero participants analyzed | 2.01 [1.69 to 2.39] | 2.17 [1.79 to 2.39] | 2.56 [2.15 to 3.05] | 2.11 [1.77 to 2.5] | 2.41 [2.01 to 2.89] | 2 [1.66 to 2.4] | NA [NA to NA] — Zero participants analyzed
  MenA 60mths N=33,35,18,31,42,27,25,23,25,23,24,30 | 2.6 [2.12 to 3.19] | 2.69 [2.21 to 3.28] | 2.85 [2.16 to 3.75] | 2.11 [1.71 to 2.61] | 2 [1.67 to 2.39] | 2.08 [1.77 to 2.45] | 2 [1.69 to 2.36] | 2.37 [1.99 to 2.82] | 2.2 [1.86 to 2.6] | 2.36 [1.98 to 2.8] | 2 [1.69 to 2.37] | 2.24 [1.91 to 2.62]
  MenC 40mths N=32,36,17,33,0,20,22,26,26,24,24,0 | 6.43 [3.85 to 11] | 7.02 [4.33 to 11] | 23 [11 to 46] | 4.29 [2.59 to 7.11] | NA [NA to NA] — Zero participants analyzed | 3.18 [1.98 to 5.1] | 2.68 [1.71 to 4.2] | 4.17 [2.77 to 6.27] | 5.45 [3.62 to 8.2] | 4.98 [3.26 to 7.62] | 6.45 [4.22 to 9.86] | NA [NA to NA] — Zero participants analyzed
  MenC 60mths N=32,34,17,31,42,21,24,22,21,22,24,30 | 4.98 [3.28 to 7.55] | 4.69 [3.13 to 7.04] | 14 [8.15 to 26] | 6.77 [4.43 to 10] | 3.93 [2.73 to 5.65] | 2.75 [1.77 to 4.26] | 2.86 [1.9 to 4.3] | 3.22 [2.11 to 4.92] | 4.02 [2.6 to 6.21] | 4.85 [3.17 to 7.4] | 6.27 [4.18 to 9.41] | 9.46 [6.48 to 14]
  MenW 40mths N=33,37,17,34,0,28,23,27,28,25,24,0 | 23 [13 to 42] | 27 [15 to 47] | 22 [9.65 to 50] | 26 [14 to 46] | NA [NA to NA] — Zero participants analyzed | 3.86 [2.15 to 6.93] | 6.77 [3.55 to 13] | 12 [6.72 to 22] | 7.55 [4.22 to 14] | 23 [13 to 43] | 16 [8.63 to 30] | NA [NA to NA] — Zero participants analyzed
  MenW 60mths N=32,34,18,31,42,26,25,23,24,21,24,30 | 18 [10 to 32] | 35 [20 to 60] | 34 [16 to 72] | 26 [15 to 45] | 6.51 [3.99 to 11] | 3.77 [2.14 to 6.64] | 7.26 [4.08 to 13] | 10 [5.77 to 19] | 7.02 [3.9 to 13] | 24 [13 to 45] | 19 [11 to 35] | 5.02 [2.88 to 8.73]
  MenY 40mths N=33,37,17,34,0,28,23,27,28,25,24,0 | 22 [13 to 38] | 15 [9.16 to 26] | 27 [13 to 58] | 9.33 [5.48 to 16] | NA [NA to NA] — Zero participants analyzed | 5.54 [3.39 to 9.06] | 4.3 [2.49 to 7.4] | 7.41 [4.5 to 12] | 3.96 [2.42 to 6.46] | 13 [7.47 to 21] | 11 [6.2 to 18] | NA [NA to NA] — Zero participants analyzed
  MenY 60mths N=33,34,17,31,42,28,25,23,23,21,23,30 | 11 [6.87 to 18] | 17 [10 to 27] | 16 [8.03 to 32] | 7.24 [4.35 to 12] | 4.36 [2.81 to 6.75] | 5.24 [3.32 to 8.27] | 4.49 [2.79 to 7.22] | 6.44 [3.94 to 11] | 3.73 [2.27 to 6.12] | 11 [6.57 to 18] | 11 [6.88 to 18] | 2.82 [1.8 to 4.42]

ADVERSE EVENTS:
Time Frame: Approximately 37 months overall (11 months of enrollment and 26 months of individual subject participation).
Description: The analyses for serious adverse events (SAEs) and adverse events (AEs) were done on the safety population (i.e., all subjects enrolled who received study vaccination and provided post-baseline safety data).
Arm/Group | UK2,3,4,12+ | UK2,4,12+ | UK2,4C/12+ | UK2,4,12- | UK Control | Ca2,4,6+ | Ca2,4,6+/12PS | Ca2,4,12+ | Ca2,4+/12PS | Ca2,4,12- | Ca2,4-/12PS | Ca Control
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/33 | 0/16 | 3/29 | 0/26 | 1/28 | 0/25 | 0/24 | 0/26 | 0/22 | 1/25 | 0/23
Other Adverse Events (participants affected / at risk) | 5/33 | 3/33 | 3/16 | 2/29 | 0/26 | 1/28 | 1/25 | 3/24 | 1/26 | 2/22 | 1/25 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UK2,3,4,12+ (N=33) | UK2,4,12+ (N=33) | UK2,4C/12+ (N=16) | UK2,4,12- (N=29) | UK Control (N=26) | Ca2,4,6+ (N=28) | Ca2,4,6+/12PS (N=25) | Ca2,4,12+ (N=24) | Ca2,4+/12PS (N=26) | Ca2,4,12- (N=22) | Ca2,4-/12PS (N=25) | Ca Control (N=23)
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asperger's disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UK2,3,4,12+ (N=33) | UK2,4,12+ (N=33) | UK2,4C/12+ (N=16) | UK2,4,12- (N=29) | UK Control (N=26) | Ca2,4,6+ (N=28) | Ca2,4,6+/12PS (N=25) | Ca2,4,12+ (N=24) | Ca2,4+/12PS (N=26) | Ca2,4,12- (N=22) | Ca2,4-/12PS (N=25) | Ca Control (N=23)
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days